CLINICAL TRIAL: NCT00139776
Title: Double-Blind Parallel-Group Randomized Study Of Efficacy And Safety Of "Continuous Use" Of Celecoxib Vs. The "Usual Use" Of Celecoxib In The Treatment Of Subjects With Chronic Osteoarthritis Of The Hip Or Knee Who Require an Anti-inflammatory Medication for Control Of Their Pain
Brief Title: Study Of "Continuous Use" Of Celecoxib Vs. "Usual or Intermittent Use"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3191173
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Results first posted 2009-05-19 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Chronic treatment osteoarthritis, Celecoxib, Continuous Use, Intermittent Use
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib - Continuous use (Active Comparator)
  Interventions: Drug: Celecoxib
- Celecoxib - Intermittent use (Active Comparator)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — 24 weeks of study treatment: 2 weeks open-label celecoxib 200 mg daily followed by 22 weeks of randomized double blind celecoxib 200 mg daily.
  Placebo used as flare medication when directed.
  Arms: Celecoxib - Continuous use
Drug: Celecoxib — 24 weeks of study treatment: 2 weeks open-label celecoxib 200 mg daily followed by 22 weeks of randomized double blind placebo daily.
  Usual or intermittent use of celecoxib 200 mg daily as flare medication when directed.
  Arms: Celecoxib - Intermittent use

SUMMARY:
To determine whether "continuous use" of celecoxib over a 6-month period is more efficacious than "usual or intermittent use" in preventing spontaneous osteoarthritis flares of the knee and hip.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed, according to American College of Rheumatology guidelines, with osteoarthritis of the hip or knee and requires non-steroidal anti-inflammatory drugs (NSAIDs) to control their osteoarthritis pain and have access to a touch-tone telephone.

Exclusion Criteria:

* Subject has had surgery on index joint.
* Subject has history of rheumatoid arthritis or fibromyalgia syndrome.
* Subject has active gastrointestinal or cardiovascular disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (115):
- United States (61):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Stockton, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, New Milford, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Clinton, Maryland
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Greenbelt, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, Manlius, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Zanesville, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Yakima, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Belgium (2):
  - Pfizer Investigational Site, Ham
  - Pfizer Investigational Site, Liège
- Brazil (3):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (19):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, North York, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Charlottetown, Prince Edward Island
  - Pfizer Investigational Site, Montague, Prince Edward Island
  - Pfizer Investigational Site, Mirabel, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Rimouski, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Ste-Foy, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Chile (3):
  - Pfizer Investigational Site, Viña del Mar, Región de Valparaíso
  - Pfizer Investigational Site, Rancagua, Región del Libertador General Bernardo O’Higgins
  - Pfizer Investigational Site, Santiago, RM
- Colombia (4):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Barranquila
  - Pfizer Investigational Site, Bogotá
  - Pfizer Investigational Site, Bucaramanga
- France (4):
  - Pfizer Investigational Site, Joué-lès-Tours
  - Pfizer Investigational Site, L'Union
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Tours
- United Kingdom (19):
  - Pfizer Investigational Site, Randalstown, Co Antrim
  - Pfizer Investigational Site, Newtownabbey, Co.Antrim
  - Pfizer Investigational Site, Leslie, Fife
  - Pfizer Investigational Site, Watford, Herts
  - Pfizer Investigational Site, Canterbury, Kent
  - Pfizer Investigational Site, Wigan, Lancs
  - Pfizer Investigational Site, Bradwell Common, Milton Keynes
  - Pfizer Investigational Site, Greenisland, Carrickfergus, Northern Ireland
  - Pfizer Investigational Site, Barry, Vale Of Glamorgan
  - Pfizer Investigational Site, Pound Hill, Crawley, West Sussex
  - Pfizer Investigational Site, Bradford-on-Avon, Wiltshire
  - Pfizer Investigational Site, Midsomer Norton, Wiltshire
  - Pfizer Investigational Site, Bangor
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Blackpool
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Cookstown
  - Pfizer Investigational Site, Trowbridge

REFERENCES:
- [Derived] Strand V, Simon LS, Dougados M, Sands GH, Bhadra P, Breazna A, Immitt J. Treatment of osteoarthritis with continuous versus intermittent celecoxib. J Rheumatol. 2011 Dec;38(12):2625-34. doi: 10.3899/jrheum.110636. Epub 2011 Nov 1. PMID 22045833
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191173&StudyName=Study%20Of%20%22Continuous%20Use%22%20Of%20Celecoxib%20Vs.%20%22Usual%20or%20Intermittent%20Use%22%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 111 centers in the Americas and Europe enrolled and treated subjects (2 centers in Belgium, 4 centers in Brazil, 20 centers in Canada, 5 centers in Chile, 5 centers in Columbia, 1 center in France, 15 centers in the United Kingdom, and 59 centers in the United States).
Pre-assignment Details: 17 participants completed Open-label run-in Period II and were randomized to Period III Double Blind but not treated.
Groups:
- Wash-Out: Discontinue Non-Steroidal Anti-Inflammatories: Period I (14+/-2 days) wash out and discontinuation of non-steroidal anti-inflammatories (NSAIDs) leading to osteoarthritis (OA) flare.
- Open-Label Celecoxib Run-in Period: Period II (14+/-2 days) run-in treatment with open label celecoxib to observe successful treatment of flare. Participants successfully treated randomized to 2 treatment groups in Period III (overall study).
- Celecoxib 200mg Continuous Use: Period III Double blind single dose of celecoxib 200 mg daily. Placebo used as flare medication when directed.
- Celecoxib 200mg Intermittent Use: Period III Double blind placebo was taken once daily. Usual or intermittent use of celecoxib 200 mg daily as flare medication when directed.
Period: Period I
Arm/Group | Wash-Out: Discontinue Non-Steroidal Anti-Inflammatories | Open-Label Celecoxib Run-in Period | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Started | 1772 | 0 | 0 | 0
Completed | 1197 | 0 | 0 | 0
Not Completed | 575 | 0 | 0 | 0
Not completed — Did not enter Period II | 575 | 0 | 0 | 0
Period: Period II
Arm/Group | Wash-Out: Discontinue Non-Steroidal Anti-Inflammatories | Open-Label Celecoxib Run-in Period | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Started | 0 | 1197 | 0 | 0
Completed | 0 | 875 | 0 | 0
Not Completed | 0 | 322 | 0 | 0
Not completed — Not Randomized into Period III | 0 | 322 | 0 | 0
Period: Period III
Arm/Group | Wash-Out: Discontinue Non-Steroidal Anti-Inflammatories | Open-Label Celecoxib Run-in Period | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Started | 0 | 0 | 431 (Randomized 440: 9 participants not treated) | 427 (Randomized 435: 8 participants not treated)
Completed | 0 | 0 | 355 | 321
Not Completed | 0 | 0 | 76 | 106
Not completed — Adverse Event | 0 | 0 | 22 | 23
Not completed — Other | 0 | 0 | 23 | 34
Not completed — Lack of Efficacy | 0 | 0 | 10 | 24
Not completed — Lost to Follow-up | 0 | 0 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 16 | 21

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib 200mg Continuous Use: Double blind single dose of celecoxib 200 mg daily. Placebo used as flare medication when directed.
- Celecoxib 200mg Intermittent Use: Double blind placebo was taken once daily. Usual or intermittent use of celecoxib 200 mg daily as flare medication when directed.
- Total: Total of all reporting groups
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use | Total
Number analyzed (Participants) | 431 | 427 | 858
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.00) | 58.7 (9.6) | 58.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 317 | 303 | 620
  Male | 114 | 124 | 238

OUTCOME MEASURES:

1. Primary Outcome: Number of Flare Events Per Time of Exposure to Study Medication
Description: Number of flare events per month during Period III (calculated as number of flares divided by number of months participant was enrolled during Period III). Flare was determined using pre-defined criteria, using an interactive voice response system.
Time Frame: Period III (22 weeks)
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication
Measure: Mean (Standard Deviation); unit: flare events per month
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
flare events per month | 0.54 (0.74) | 0.93 (1.01)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Null hypothesis for primary outcome is that there is no difference in the number of flares observed between the 2 treatment arms of celecoxib 200mg continuous use and celecoxib 200mg intermittent use. Sample size calculation: Sufficient number of participants were randomized to provide at least 80% power to detect an estimated effect size of 0.2 using a 2-sided t-test at a 0.05 significant level; Test type: Superiority or Other; p < 0.0001, ANOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect

2. Secondary Outcome: Time to Occurrence of First Osteoarthritis (OA) Flare
Description: Time from first dose of double blind medication (start of Period III) to occurrence of first OA flare. Flare was determined using pre-defined criteria, using an interactive voice response system
Time Frame: Period III (22 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
days | 16.0 [14.0 to 22.0] | 8.0 [8.0 to 9.0]
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Kaplan-Meier analysis; Test type: Superiority or Other; p < 0.0001, Log Rank — Threshold for statistical significance p<0.05

3. Secondary Outcome: Proportion of Days Free From Osteoarthritis (OA) Flare
Description: Number of days subject was free from OA flare divided by number of days on study medication in Period III. Flare was determined using pre-defined criteria, using an interactive voice response system.
Time Frame: Period III (22 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of days free from OA flare
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
proportion of days free from OA flare | 0.77 (0.28) | 0.67 (0.30)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Test type: Superiority or Other; p < 0.0001, ANOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect

4. Secondary Outcome: Proportion of Days in Osteoarthritis (OA) Flare
Description: Number of days subject was in OA flare divided by number of days on study medication in Period III. Subjects may have more than one flare. Flare was determined using pre-defined criteria, using an interactive voice response system.
Time Frame: Period III (22 weeks)
Measure: Mean (Standard Deviation); unit: proportion of days in OA flare
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
proportion of days in OA flare | 0.23 (0.28) | 0.33 (0.30)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Test type: Superiority or Other; p < 0.0001, ANOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect

5. Secondary Outcome: Arthritis Pain Numerical Rating Scale (NRS)
Description: Participant rated intensity of osteoarthritis pain on categorical scale from 0 (no pain) to 10 (worst pain). Scores analyzed as area under the curve (AUC) of participant's scores from each assessment in Period III.
Time Frame: Period III
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication.
  These data are presented by the weeks from the start of Period II, 2 weeks before randomization. The weeks post-randomization, Period III, are different from the study weeks i.e. includes 2 weeks from Period II.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale * weeks
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
scores on a scale * weeks
  Week 4 (n=415 cont; n=414 inter) | 81.7 (1.1) | 90.5 (1.1)
  Week 8 (n=401 cont; n=395 inter) | 148.8 (2.6) | 167.0 (2.6)
  Week 12 (n=383 cont; n=363 inter) | 212.6 (4.1) | 234.3 (4.1)
  Week 16 (n=373 cont; n=339 inter) | 272.7 (5.9) | 297.6 (5.9)
  Week 20 (n=362; n=323 inter) | 335.9 (7.8) | 361.1 (7.8)
  Week 24 (n=350 cont; n=403 inter) | 378.1 (9.1) | 403.9 (9.2)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 8; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 3: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 12; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 4: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 16; Test type: Superiority or Other; p = 0.003, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 5: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 20; Test type: Superiority or Other; p = 0.022, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 6: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 24; Test type: Superiority or Other; p = 0.047, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate

6. Secondary Outcome: Patient's Global Assessment of Arthritis
Description: Participant's response to question "Considering all the ways the osteoarthritis in your hip or knee affects you, how are you doing today?" on scale from 1 (very good) to 5 (very poor). Scores analyzed as area under the curve (AUC) of participant's scores from each assessment in Period III.
Time Frame: Period III
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: scores on a scale * weeks
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
scores on a scale * weeks
  Week 4 (n=415 cont; n=414 inter) | 67.9 (0.68) | 71.7 (0.69)
  Week 8 (n=401 cont; n=395 inter) | 126.0 (1.55) | 133.2 (1.56)
  Week 12 (n=383 cont; n=363 inter) | 182.8 (2.48) | 188.7 (2.48)
  Week 16 (n=373 cont; n=339 inter) | 236.3 (3.59) | 241.2 (3.59)
  Week 20 (n=362 cont; n=323 inter) | 292.4 (4.83) | 293.8 (4.84)
  Week 24 (n=350 cont; n=309 inter) | 329.2 (5.75) | 328.9 (5.76)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 8; Test type: Superiority or Other; p = 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 3: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 12; Test type: Superiority or Other; p = 0.096, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 4: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 16; Test type: Superiority or Other; p = 0.338, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 5: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 20; Test type: Superiority or Other; p = 0.832, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 6: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Week 24; Test type: Superiority or Other; p = 0.972, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate

7. Secondary Outcome: Physician's Global Assessment of Arthritis at Final Visit
Description: Physician assessed each participant's disease symptoms on a categorical scale from 1 (very good) to 5 (very poor).
Time Frame: Period III (22 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
participants
  Grade 1 (very good) | 68 | 39
  Grade 2 (good) | 242 | 244
  Grade 3 (fair) | 91 | 113
  Grade 4 (poor) | 23 | 27
  Grade 5 (very poor) | 2 | 2
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Test type: Superiority or Other; p = 0.0046, Cochran-Mantel-Haenszel — Overall p-value Threshold for statistical significance p<0.05; Test of row mean score differences based on modified ridits (standardizing the mid-rank)

8. Secondary Outcome: Total Rescue Medication Taken (Mean)
Description: Total amount of rescue medication (acetaminophen in milligrams [mg]) taken per month per participant
Time Frame: Period III (22 weeks)
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication.
  Subjects who did not take rescue medication were assumed to have taken 0mg and were included in the analysis.
  Number of subjects taking rescue medication: continuous use n=220; intermittent use n=239.
Measure: Mean (Standard Deviation); unit: mg taken per month per participant
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
mg taken per month per participant | 1566 (4840) | 2428 (4974)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Test type: Superiority or Other; p = 0.0102, ANOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect

9. Secondary Outcome: Proportion of Days on Rescue Medication
Description: Days on rescue medication divided by number of days on study medication in Period III
Time Frame: Period III (22 weeks)
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication. Number of subjects taking rescue medication: continuous use n=220; intermittent use n=239.
  Subjects who did not take rescue medication were calculated as 0 and included in the analysis.
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
proportion of days | 0.044 (0.102) | 0.069 (0.121)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Test type: Superiority or Other; p = 0.0012, ANOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect

10. Secondary Outcome: Days on Flare Medication
Description: Number of days on flare medication per month per subject calculated as number of days on flare medication divided by the number of days on study medication in Period III
Time Frame: Period III (22 weeks)
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication.
  Subjects who did not take flare medication were calculated as 0 and included in the analysis.
  Number of subjects taking flare medication: continuous use n=282; intermittent use n=339.
Measure: Mean (Standard Deviation); unit: days on medication per month per subject
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
days on medication per month per subject | 6.589 (8.589) | 9.793 (9.253)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Test type: Superiority or Other; p < 0.0001, ANOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect

11. Secondary Outcome: Change in Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Scores
Description: Score at end of Period III minus score at start of Period III. WOMAC assesses subject responses to 24 components regarding subscales of pain, stiffness and physical function (score range: 0=none to 4= extreme). Total score is sum of the 3 subscale scores. Negative change indicates improvement.
Time Frame: Period III (22 weeks)
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication. Number of subjects evaluable: continuous use Period III start n=428, end n=427; intermittent use Period III start n=424, end n=424
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
scores on a scale
  Total WOMAC score | 1.60 (0.71) | 4.99 (0.71)
  WOMAC pain subscale | 0.37 (0.15) | 1.18 (0.15)
  WOMAC stiffness subscale | 0.12 (0.07) | 0.40 (0.07)
  WOMAC physical function subscale | 1.13 (0.51) | 3.43 (0.51)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Total WOMAC score; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Celecoxib 200mg Continuous Use; Total WOMAC score - Continuous use; Test type: Superiority or Other; Mean Difference (Final Values) = 1.60, 95% CI [0.21 to 2.99], Standard Error of Mean 0.71 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 3: Comparison: Celecoxib 200mg Intermittent Use; Total WOMAC score - Intermittent use; Test type: Superiority or Other; Mean Difference (Final Values) = 4.99, 95% CI [3.60 to 6.38], Standard Error of Mean 0.71 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 4: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC pain subscale; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 5: Comparison: Celecoxib 200mg Continuous Use; WOMAC pain subscale - Continuous use; Test type: Superiority or Other; Mean Difference (Final Values) = 0.37, 95% CI [0.06 to 0.67], Standard Error of Mean 0.15 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 6: Comparison: Celecoxib 200mg Intermittent Use; WOMAC pain subscale - Intermittent use; Test type: Superiority or Other; Mean Difference (Final Values) = 1.18, 95% CI [0.88 to 1.49], Standard Error of Mean 0.15 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 7: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC stiffness subscale; Test type: Superiority or Other; p = 0.004, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 8: Comparison: Celecoxib 200mg Continuous Use; WOMAC stiffness subscale - Continuous use; Test type: Superiority or Other; Mean Difference (Final Values) = 0.12, 95% CI [-0.02 to 0.25], Standard Error of Mean 0.07 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 9: Comparison: Celecoxib 200mg Intermittent Use; WOMAC stiffness subscale - Intermittent use; Test type: Superiority or Other; Mean Difference (Final Values) = 0.40, 95% CI [0.26 to 0.53], Standard Error of Mean 0.07 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 10: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC physical function subscale; Test type: Superiority or Other; p = 0.002, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 11: Comparison: Celecoxib 200mg Continuous Use; WOMAC physical function subscale - Continuous use; Test type: Superiority or Other; Mean Difference (Final Values) = 1.13, 95% CI [0.13 to 2.14], Standard Error of Mean 0.51 — Change in LSmean (score at end of Period III minus score at start of Period III)
Statistical Analysis 12: Comparison: Celecoxib 200mg Intermittent Use; WOMAC physical function subscale - Intermittent use; Test type: Superiority or Other; Mean Difference (Final Values) = 3.43, 95% CI [2.42 to 4.43], Standard Error of Mean 0.51 — Change in LSmean (score at end of Period III minus score at start of Period III)

12. Other Pre Specified Outcome: Change in Medical Outcomes Study Sleep Scale - All Assessments
Description: Subject assessment on 7 sleep associated categories. Raw scores are transformed to a 0-100 scale. Higher score indicates more of the outcome (e.g. more snoring, more adequate sleep). Score at end of Period III minus score at start of Period III.
Time Frame: Period III
Population: Intent to treat (ITT) population included subjects who were randomized and received at least one dose of double blind study medication. Subjects assessed per scale n=continuous use (cont); n=intermittent use (inter)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
scores on a scale
  Sleep disturbance (n=415 cont; n=410 inter) | 0.5 (15.95) | -1.4 (15.55)
  Snoring (n=415 cont; n=412 inter) | 0.9 (22.36) | 0.7 (21.73)
  Awaken short of breath (n=417 cont; n=411 inter) | 1.9 (16.14) | 1.1 (20.00)
  Quantity of sleep (n=417 cont; n=413 inter) | -0.1 (0.91) | -0.1 (0.89)
  Sleep adequacy (n=416 cont; n=413 inter) | 0.1 (24.47) | -1.3 (22.26)
  Somnolence (n=416 cont; n=413 inter) | 1.4 (14.55) | 0.6 (13.70)
  Sleep problems index I (n=416 cont; n=410 inter) | 0.9 (13.20) | 0.5 (13.18)
  Sleep problems index II (n=413 cont; n=408 inter) | 0.7 (12.29) | -0.1 (12.14)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Sleep disturbance; Test type: Superiority or Other; p = 0.2712, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Snoring; Test type: Superiority or Other; p = 0.8737, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 3: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Awaken short of breath; Test type: Superiority or Other; p = 0.7703, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 4: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Quantity of sleep; Test type: Superiority or Other; p = 0.3769, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 5: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Sleep adequacy; Test type: Superiority or Other; p = 0.4075, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 6: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Somnolence; Test type: Superiority or Other; p = 0.5854, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 7: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Sleep problems index I; Test type: Superiority or Other; p = 0.8358, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 8: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Sleep problems index II; Test type: Superiority or Other; p = 0.5878, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate

13. Secondary Outcome: Area Under the Curve (AUCs) of Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Scores
Description: WOMAC assesses subject responses to 24 components regarding subscales of pain, stiffness and physical function (score range: 0=none to 4= extreme). Total score is sum of the 3 subscale scores. Scores analyzed as area under the curve (AUC) of participant's WOMAC scores from each assessment in Period III.
Time Frame: Period III (22 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: scores on a scale * weeks
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
scores on a scale * weeks
  Total WOMAC score | 604.9 (313.10) | 693.6 (317.30)
  WOMAC pain subscale | 119.2 (63.36) | 138.4 (65.95)
  WOMAC stiffness subscale | 54.5 (27.57) | 62.1 (27.7)
  WOMAC physical function subscale | 431.4 (229.38) | 493.6 (230.74)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC total score; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC pain subscale; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 3: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC stiffness subscale; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 4: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; WOMAC physical function subscale; Test type: Superiority or Other; p < 0.001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate

14. Other Pre Specified Outcome: Medical Outcomes Study Sleep Scale - Number of Participants With Optimal, Mixed and Not Optimal Sleep
Description: Transformed score scale: 1=optimal; 0=not optimal; mixed = both optimal and non-optimal sleep during Period III
Time Frame: Period III
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
participants
  Optimal (all scores are 1) | 139 | 123
  Mixed (scores are both 1 and 0) | 166 | 165
  Not optimal (all scores are 0) | 115 | 132
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Analysis across all 3 sleep scores for Period III; Test type: Superiority or Other; p = 0.1437, Cochran-Mantel-Haenszel — Threshold for statistical significance p<0.05; by general association

15. Other Pre Specified Outcome: Change in the Quality of Life Short Form-12v2 (SF-12v2) Scale Scores - All Assessments
Description: SF-12v2 is a 12 item health survey covering 7 topics. Raw scores are transformed to a 0 to 100 scale. Higher scores indicate better state of health. Score at end of Period III minus score at start of Period III.
Time Frame: Period III
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Number analyzed (Participants) | 431 | 427
scores on a scale
  Physical function (n=417 cont; n=413 inter) | 1.8 (23.03) | -3.2 (22.77)
  Role physical (n=416 cont; n=412 inter) | 3.5 (19.93) | -1.1 (20.07)
  Bodily pain (n=417 cont; n=414 inter) | 3.8 (20.11) | -0.3 (21.56)
  General health (n=417 cont; n=414 inter) | -0.3 (17.60) | -0.8 (17.27)
  Vitality (n=416 cont; n=414 inter) | 0.3 (20.43) | -3.5 (18.34)
  Social functioning (n=416 cont; n=414 inter) | -1.9 (20.16) | -3.5 (22.37)
  Role emotional (n=417 cont; n=413 inter) | -0.7 (18.62) | -2.1 (19.80)
  Mental health (n=416 cont; n=413 inter) | -0.9 (15.57) | -1.3 (16.05)
  Physical component summary(n=416 cont;n=411 inter) | 9.0 (55.55) | -5.2 (57.48)
  Mental component summary (n=416 cont;n=411 inter) | -3.1 (51.59) | -10.5 (55.66)
Statistical Analysis 1: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Physical function; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 2: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Role physical; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 3: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Bodily pain; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 4: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; General health; Test type: Superiority or Other; p = 0.3097, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 5: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Vitality; Test type: Superiority or Other; p = 0.0139, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 6: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Social functioning; Test type: Superiority or Other; p = 0.1303, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 7: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Role emotional; Test type: Superiority or Other; p = 0.1404, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 8: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Mental health; Test type: Superiority or Other; p = 0.4015, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 9: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Physical component summary; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate
Statistical Analysis 10: Comparison: Celecoxib 200mg Continuous Use vs Celecoxib 200mg Intermittent Use; Mental component summary; Test type: Superiority or Other; p = 0.0301, ANCOVA — Threshold for statistical significance p<0.05; Treatment as fixed effect and baseline as covariate

16. Other Pre Specified Outcome: Serious Adverse Events in Open Label run-in Period
Description: Serious adverse events occuring during the 2 week run-in period (Period II) when all participants were dosed with celecoxib 200 mg daily
Time Frame: 2 weeks prior to double blind dosing
Population: 1197 participants entered the open-label run-in (period II) to allow observation of successful treatment of an osteoarthritis flare. 875 participants were randomized to double blind treatment (period III). 322 participants were not randomized.
Measure: Number; unit: participants
Groups:
- Celecoxib 200mg Open Label: Period II run-in (2 weeks). Celecoxib 200 mg daily until resolution of screening osteoarthritis flare as defined by IVRS
Arm/Group | Celecoxib 200mg Open Label
Number analyzed (Participants) | 1197
participants
  Anaemia | 1
  Vitreous haemorrhage | 1

ADVERSE EVENTS:
Arm/Group | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Serious Adverse Events (participants affected / at risk) | 6 | 10
Other Adverse Events (participants affected / at risk) | 242 | 246
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Atrial fibrillation (Cardiac disorders) | 1/431 | 0/427
Coronary artery disease (Cardiac disorders) | 1/431 | 0/427
Abdominal pain (Gastrointestinal disorders) | 0/431 | 1/427
Gastritis (Gastrointestinal disorders) | 0/431 | 1/427
Melaena (Gastrointestinal disorders) | 1/431 | 0/427
Pancreatitis (Gastrointestinal disorders) | 0/431 | 1/427
Rectal haemorrhage (Gastrointestinal disorders) | 1/431 | 0/427
Chest pain (General disorders) | 1/431 | 1/427
Non-cardiac chest pain (General disorders) | 0/431 | 1/427
Skin laceration (Injury, poisoning and procedural complications) | 0/431 | 1/427
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/431 | 0/427
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/431 | 1/427
Transient ischaemic attack (Nervous system disorders) | 0/431 | 1/427
Bipolar I disorder (Psychiatric disorders) | 0/431 | 1/427
Nephrolithiasis (Renal and urinary disorders) | 1/431 | 0/427
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/431 | 0/427
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/431 | 0/427
Knee arthroplasty (Surgical and medical procedures) | 0/431 | 1/427
Hypertensive crisis (Vascular disorders) | 0/431 | 1/427
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Celecoxib 200mg Continuous Use | Celecoxib 200mg Intermittent Use
Anaemia (Blood and lymphatic system disorders) | 1/431 | 0/427
Lymphadenopathy (Blood and lymphatic system disorders) | 1/431 | 2/427
Angina pectoris (Cardiac disorders) | 1/431 | 0/427
Bundle branch block left (Cardiac disorders) | 1/431 | 0/427
Extrasystoles (Cardiac disorders) | 1/431 | 0/427
Hypertensive heart disease (Cardiac disorders) | 0/431 | 1/427
Sinus tachycardia (Cardiac disorders) | 0/431 | 1/427
Tachycardia (Cardiac disorders) | 1/431 | 0/427
Cerumen impaction (Ear and labyrinth disorders) | 1/431 | 1/427
Deafness (Ear and labyrinth disorders) | 1/431 | 0/427
Ear disorder (Ear and labyrinth disorders) | 1/431 | 0/427
Ear pain (Ear and labyrinth disorders) | 2/431 | 2/427
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0/431 | 1/427
Tympanic membrane disorder (Ear and labyrinth disorders) | 1/431 | 0/427
Vertigo (Ear and labyrinth disorders) | 5/431 | 3/427
Goitre (Endocrine disorders) | 1/431 | 0/427
Hypothyroidism (Endocrine disorders) | 0/431 | 1/427
Cataract (Eye disorders) | 0/431 | 1/427
Conjunctivitis (Eye disorders) | 1/431 | 0/427
Conjunctivitis allergic (Eye disorders) | 1/431 | 0/427
Diplopia (Eye disorders) | 1/431 | 0/427
Dry eye (Eye disorders) | 2/431 | 0/427
Eye allergy (Eye disorders) | 1/431 | 0/427
Eye irritation (Eye disorders) | 0/431 | 1/427
Glaucoma (Eye disorders) | 1/431 | 0/427
Lacrimation increased (Eye disorders) | 1/431 | 1/427
Myodesopsia (Eye disorders) | 0/431 | 1/427
Vision blurred (Eye disorders) | 2/431 | 1/427
Visual acuity reduced (Eye disorders) | 1/431 | 0/427
Abdominal discomfort (Gastrointestinal disorders) | 1/431 | 1/427
Abdominal distension (Gastrointestinal disorders) | 3/431 | 1/427
Abdominal hernia (Gastrointestinal disorders) | 1/431 | 0/427
Abdominal pain (Gastrointestinal disorders) | 10/431 | 3/427
Abdominal pain lower (Gastrointestinal disorders) | 1/431 | 0/427
Abdominal pain upper (Gastrointestinal disorders) | 7/431 | 10/427
Aphthous stomatitis (Gastrointestinal disorders) | 1/431 | 0/427
Breath odour (Gastrointestinal disorders) | 0/431 | 1/427
Colitis (Gastrointestinal disorders) | 1/431 | 2/427
Constipation (Gastrointestinal disorders) | 5/431 | 4/427
Dental caries (Gastrointestinal disorders) | 0/431 | 1/427
Diarrhoea (Gastrointestinal disorders) | 7/431 | 17/427
Dry mouth (Gastrointestinal disorders) | 1/431 | 0/427
Dyspepsia (Gastrointestinal disorders) | 17/431 | 6/427
Eructation (Gastrointestinal disorders) | 0/431 | 1/427
Flatulence (Gastrointestinal disorders) | 2/431 | 0/427
Frequent bowel movements (Gastrointestinal disorders) | 1/431 | 0/427
Gastritis (Gastrointestinal disorders) | 5/431 | 2/427
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4/431 | 3/427
Gastrooesophagitis (Gastrointestinal disorders) | 1/431 | 0/427
Gingival pain (Gastrointestinal disorders) | 1/431 | 1/427
Haematochezia (Gastrointestinal disorders) | 0/431 | 1/427
Haemorrhoids (Gastrointestinal disorders) | 1/431 | 1/427
Inguinal hernia (Gastrointestinal disorders) | 0/431 | 1/427
Irritable bowel syndrome (Gastrointestinal disorders) | 3/431 | 3/427
Mouth ulceration (Gastrointestinal disorders) | 1/431 | 0/427
Nausea (Gastrointestinal disorders) | 5/431 | 9/427
Oral pain (Gastrointestinal disorders) | 0/431 | 1/427
Paraesthesia oral (Gastrointestinal disorders) | 1/431 | 0/427
Parotid gland enlargement (Gastrointestinal disorders) | 0/431 | 1/427
Peptic ulcer (Gastrointestinal disorders) | 1/431 | 0/427
Proctitis (Gastrointestinal disorders) | 0/431 | 1/427
Rectal haemorrhage (Gastrointestinal disorders) | 1/431 | 1/427
Stomach discomfort (Gastrointestinal disorders) | 4/431 | 1/427
Stomatitis (Gastrointestinal disorders) | 1/431 | 0/427
Tongue disorder (Gastrointestinal disorders) | 0/431 | 1/427
Toothache (Gastrointestinal disorders) | 3/431 | 6/427
Vomiting (Gastrointestinal disorders) | 5/431 | 6/427
Asthenia (General disorders) | 1/431 | 0/427
Chest discomfort (General disorders) | 1/431 | 0/427
Chest pain (General disorders) | 2/431 | 4/427
Fatigue (General disorders) | 6/431 | 9/427
Feeling hot (General disorders) | 0/431 | 1/427
Gravitational oedema (General disorders) | 0/431 | 1/427
Hypothermia (General disorders) | 0/431 | 1/427
Influenza like illness (General disorders) | 1/431 | 4/427
Malaise (General disorders) | 0/431 | 1/427
Oedema peripheral (General disorders) | 4/431 | 12/427
Pain (General disorders) | 6/431 | 9/427
Pyrexia (General disorders) | 2/431 | 5/427
Swelling (General disorders) | 0/431 | 1/427
Thirst (General disorders) | 0/431 | 1/427
Cholelithiasis (Hepatobiliary disorders) | 1/431 | 0/427
Hypersensitivity (Immune system disorders) | 0/431 | 1/427
Seasonal allergy (Immune system disorders) | 2/431 | 1/427
Alveolar osteitis (Infections and infestations) | 0/431 | 1/427
American trypanosomiasis (Infections and infestations) | 0/431 | 1/427
Amoebiasis (Infections and infestations) | 0/431 | 1/427
Bronchitis (Infections and infestations) | 4/431 | 9/427
Cellulitis (Infections and infestations) | 2/431 | 2/427
Cystitis (Infections and infestations) | 1/431 | 4/427
Diverticulitis (Infections and infestations) | 0/431 | 1/427
Ear infection (Infections and infestations) | 1/431 | 0/427
Fungal skin infection (Infections and infestations) | 0/431 | 1/427
Gastroenteritis (Infections and infestations) | 2/431 | 0/427
Gastroenteritis viral (Infections and infestations) | 1/431 | 1/427
Groin abscess (Infections and infestations) | 0/431 | 1/427
Herpes zoster (Infections and infestations) | 1/431 | 3/427
Infected bites (Infections and infestations) | 1/431 | 0/427
Influenza (Infections and infestations) | 10/431 | 9/427
Labyrinthitis (Infections and infestations) | 1/431 | 1/427
Laryngitis (Infections and infestations) | 1/431 | 0/427
Localised infection (Infections and infestations) | 2/431 | 0/427
Lower respiratory tract infection (Infections and infestations) | 1/431 | 1/427
Lymph gland infection (Infections and infestations) | 1/431 | 0/427
Nail infection (Infections and infestations) | 1/431 | 0/427
Nasopharyngitis (Infections and infestations) | 19/431 | 20/427
Onychomycosis (Infections and infestations) | 1/431 | 1/427
Oral herpes (Infections and infestations) | 1/431 | 0/427
Osteomyelitis (Infections and infestations) | 0/431 | 1/427
Otitis externa (Infections and infestations) | 1/431 | 0/427
Otitis media (Infections and infestations) | 0/431 | 1/427
Otitis media acute (Infections and infestations) | 0/431 | 1/427
Parasitic gastroenteritis (Infections and infestations) | 0/431 | 1/427
Pharyngitis (Infections and infestations) | 4/431 | 3/427
Pharyngitis streptococcal (Infections and infestations) | 1/431 | 0/427
Pyelonephritis (Infections and infestations) | 1/431 | 0/427
Pyoderma (Infections and infestations) | 1/431 | 1/427
Rhinitis (Infections and infestations) | 1/431 | 1/427
Sinusitis (Infections and infestations) | 11/431 | 10/427
Sinusitis bacterial (Infections and infestations) | 1/431 | 0/427
Tonsillitis (Infections and infestations) | 1/431 | 0/427
Tooth abscess (Infections and infestations) | 1/431 | 0/427
Tooth infection (Infections and infestations) | 0/431 | 1/427
Upper respiratory tract infection (Infections and infestations) | 14/431 | 19/427
Urinary tract infection (Infections and infestations) | 7/431 | 7/427
Viral infection (Infections and infestations) | 3/431 | 4/427
Viral pharyngitis (Infections and infestations) | 1/431 | 0/427
Viral upper respiratory tract infection (Infections and infestations) | 1/431 | 1/427
Vulvovaginal candidiasis (Infections and infestations) | 0/431 | 1/427
Vulvovaginal mycotic infection (Infections and infestations) | 0/431 | 2/427
Vulvovaginitis (Infections and infestations) | 0/431 | 1/427
Wound infection (Infections and infestations) | 0/431 | 1/427
Animal bite (Injury, poisoning and procedural complications) | 0/431 | 1/427
Arthropod bite (Injury, poisoning and procedural complications) | 1/431 | 0/427
Arthropod sting (Injury, poisoning and procedural complications) | 1/431 | 0/427
Back injury (Injury, poisoning and procedural complications) | 0/431 | 2/427
Burns second degree (Injury, poisoning and procedural complications) | 0/431 | 1/427
Contusion (Injury, poisoning and procedural complications) | 3/431 | 7/427
Device breakage (Injury, poisoning and procedural complications) | 0/431 | 1/427
Epicondylitis (Injury, poisoning and procedural complications) | 4/431 | 0/427
Excoriation (Injury, poisoning and procedural complications) | 0/431 | 2/427
Eye injury (Injury, poisoning and procedural complications) | 1/431 | 0/427
Fall (Injury, poisoning and procedural complications) | 1/431 | 2/427
Joint injury (Injury, poisoning and procedural complications) | 3/431 | 0/427
Joint sprain (Injury, poisoning and procedural complications) | 2/431 | 2/427
Limb crushing injury (Injury, poisoning and procedural complications) | 0/431 | 1/427
Limb injury (Injury, poisoning and procedural complications) | 1/431 | 0/427
Meniscus lesion (Injury, poisoning and procedural complications) | 0/431 | 1/427
Muscle injury (Injury, poisoning and procedural complications) | 1/431 | 0/427
Muscle strain (Injury, poisoning and procedural complications) | 1/431 | 2/427
Neck injury (Injury, poisoning and procedural complications) | 0/431 | 2/427
Post-traumatic pain (Injury, poisoning and procedural complications) | 1/431 | 0/427
Procedural pain (Injury, poisoning and procedural complications) | 2/431 | 0/427
Repetitive strain injury (Injury, poisoning and procedural complications) | 1/431 | 0/427
Rib fracture (Injury, poisoning and procedural complications) | 0/431 | 1/427
Skeletal injury (Injury, poisoning and procedural complications) | 1/431 | 1/427
Skin laceration (Injury, poisoning and procedural complications) | 2/431 | 0/427
Snake bite (Injury, poisoning and procedural complications) | 1/431 | 0/427
Thermal burn (Injury, poisoning and procedural complications) | 0/431 | 1/427
Tooth fracture (Injury, poisoning and procedural complications) | 1/431 | 0/427
Wrist fracture (Injury, poisoning and procedural complications) | 1/431 | 0/427
Alanine aminotransferase increased (Investigations) | 1/431 | 0/427
Aspartate aminotransferase increased (Investigations) | 1/431 | 0/427
Blood cholesterol increased (Investigations) | 0/431 | 1/427
Blood creatinine increased (Investigations) | 0/431 | 2/427
Blood potassium increased (Investigations) | 0/431 | 1/427
Blood pressure increased (Investigations) | 0/431 | 4/427
Blood urea increased (Investigations) | 0/431 | 2/427
Blood urine present (Investigations) | 0/431 | 1/427
Cardiac murmur (Investigations) | 0/431 | 1/427
Gamma-glutamyltransferase increased (Investigations) | 1/431 | 0/427
Heart rate irregular (Investigations) | 1/431 | 0/427
Hepatic enzyme increased (Investigations) | 1/431 | 0/427
Hepatitis C positive (Investigations) | 0/431 | 1/427
Weight increased (Investigations) | 1/431 | 1/427
Diabetes mellitus (Metabolism and nutrition disorders) | 1/431 | 2/427
Fluid retention (Metabolism and nutrition disorders) | 1/431 | 1/427
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1/431 | 1/427
Hyperglycaemia (Metabolism and nutrition disorders) | 1/431 | 1/427
Hyperlipdaemia (Metabolism and nutrition disorders) | 0/431 | 1/427
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1/431 | 0/427
Increased appetite (Metabolism and nutrition disorders) | 1/431 | 0/427
Polydipsia (Metabolism and nutrition disorders) | 0/431 | 1/427
Vitamin D deficiency (Metabolism and nutrition disorders) | 0/431 | 1/427
Arthralgia (Musculoskeletal and connective tissue disorders) | 17/431 | 25/427
Arthritis (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Back pain (Musculoskeletal and connective tissue disorders) | 20/431 | 31/427
Bone pain (Musculoskeletal and connective tissue disorders) | 3/431 | 0/427
Bursitis (Musculoskeletal and connective tissue disorders) | 6/431 | 2/427
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/431 | 0/427
Coccydynia (Musculoskeletal and connective tissue disorders) | 1/431 | 0/427
Costochondritis (Musculoskeletal and connective tissue disorders) | 1/431 | 0/427
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1/431 | 0/427
Flank pain (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Groin pain (Musculoskeletal and connective tissue disorders) | 1/431 | 2/427
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1/431 | 2/427
Joint swelling (Musculoskeletal and connective tissue disorders) | 1/431 | 1/427
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10/431 | 5/427
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7/431 | 12/427
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Myalgia (Musculoskeletal and connective tissue disorders) | 10/431 | 9/427
Neck pain (Musculoskeletal and connective tissue disorders) | 7/431 | 7/427
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7/431 | 2/427
Osteopenia (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18/431 | 21/427
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Periarthritis (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0/431 | 3/427
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1/431 | 0/427
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Synovitis (Musculoskeletal and connective tissue disorders) | 1/431 | 0/427
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0/431 | 1/427
Tendon pain (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Tendonitis (Musculoskeletal and connective tissue disorders) | 0/431 | 2/427
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/431 | 0/427
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/431 | 1/427
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/431 | 1/427
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/431 | 1/427
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/431 | 1/427
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/431 | 0/427
Carpal tunnel syndrome (Nervous system disorders) | 1/431 | 0/427
Cluster headache (Nervous system disorders) | 1/431 | 0/427
Dizziness (Nervous system disorders) | 8/431 | 8/427
Dysgeusia (Nervous system disorders) | 1/431 | 0/427
Facial palsy (Nervous system disorders) | 0/431 | 1/427
Headache (Nervous system disorders) | 65/431 | 68/427
Hypoaesthesia (Nervous system disorders) | 1/431 | 0/427
Lethargy (Nervous system disorders) | 1/431 | 0/427
Lumbar radiculopathy (Nervous system disorders) | 0/431 | 1/427
Migraine (Nervous system disorders) | 1/431 | 2/427
Migraine with aura (Nervous system disorders) | 1/431 | 0/427
Neuropathy peripheral (Nervous system disorders) | 1/431 | 0/427
Paraesthesia (Nervous system disorders) | 2/431 | 3/427
Poor quality sleep (Nervous system disorders) | 1/431 | 0/427
Restless legs syndrome (Nervous system disorders) | 0/431 | 1/427
Sciatica (Nervous system disorders) | 1/431 | 2/427
Sinus headache (Nervous system disorders) | 2/431 | 1/427
Somnolence (Nervous system disorders) | 1/431 | 1/427
Syncope (Nervous system disorders) | 1/431 | 0/427
Tension headache (Nervous system disorders) | 0/431 | 1/427
Tremor (Nervous system disorders) | 2/431 | 1/427
Adjustment disorder (Psychiatric disorders) | 0/431 | 1/427
Anxiety (Psychiatric disorders) | 4/431 | 1/427
Attention deficit / hyperactivity disorder (Psychiatric disorders) | 1/431 | 0/427
Confusional state (Psychiatric disorders) | 1/431 | 0/427
Depressed mood (Psychiatric disorders) | 1/431 | 0/427
Depression (Psychiatric disorders) | 5/431 | 3/427
Disorientation (Psychiatric disorders) | 0/431 | 1/427
Insomnia (Psychiatric disorders) | 11/431 | 8/427
Libido decreased (Psychiatric disorders) | 2/431 | 0/427
Nervousness (Psychiatric disorders) | 1/431 | 0/427
Nightmare (Psychiatric disorders) | 1/431 | 0/427
Restlessness (Psychiatric disorders) | 0/431 | 1/427
Sleep disorder (Psychiatric disorders) | 0/431 | 1/427
Stress (Psychiatric disorders) | 0/431 | 1/427
Dysuria (Renal and urinary disorders) | 2/431 | 0/427
Haematuria (Renal and urinary disorders) | 0/431 | 1/427
Hypertonic bladder (Renal and urinary disorders) | 1/431 | 0/427
Micturition frequency decreased (Renal and urinary disorders) | 0/431 | 1/427
Nephrolithiasis (Renal and urinary disorders) | 0/431 | 2/427
Oliguria (Renal and urinary disorders) | 0/431 | 1/427
Pollakiuria (Renal and urinary disorders) | 0/431 | 2/427
Renal colic (Renal and urinary disorders) | 0/431 | 1/427
Renal pain (Renal and urinary disorders) | 2/431 | 0/427
Urine odour abnormal (Renal and urinary disorders) | 1/431 | 0/427
Adnexa uteri pain (Reproductive system and breast disorders) | 1/431 | 0/427
Breast mass (Reproductive system and breast disorders) | 0/431 | 1/427
Breast pain (Reproductive system and breast disorders) | 1/431 | 0/427
Dysmenorrhoea (Reproductive system and breast disorders) | 2/431 | 4/427
Erectile dysfunction (Reproductive system and breast disorders) | 1/431 | 1/427
Menorrhagia (Reproductive system and breast disorders) | 0/431 | 1/427
Menstrual disorder (Reproductive system and breast disorders) | 0/431 | 1/427
Uterine polyp (Reproductive system and breast disorders) | 0/431 | 2/427
Vulvovaginal dryness (Reproductive system and breast disorders) | 0/431 | 1/427
Asthma (Respiratory, thoracic and mediastinal disorders) | 4/431 | 2/427
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Cough (Respiratory, thoracic and mediastinal disorders) | 4/431 | 4/427
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3/431 | 3/427
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/431 | 0/427
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5/431 | 3/427
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1/431 | 0/427
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7/431 | 4/427
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1/431 | 0/427
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1/431 | 1/427
Rales (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3/431 | 2/427
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2/431 | 0/427
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3/431 | 2/427
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/431 | 1/427
Alopecia (Skin and subcutaneous tissue disorders) | 2/431 | 0/427
Blister (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Dermatitis (Skin and subcutaneous tissue disorders) | 0/431 | 3/427
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/431 | 1/427
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Eczema (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Erythema (Skin and subcutaneous tissue disorders) | 2/431 | 0/427
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0/431 | 2/427
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Ingrown hair (Skin and subcutaneous tissue disorders) | 0/431 | 1/427
Pruritus (Skin and subcutaneous tissue disorders) | 3/431 | 2/427
Rash (Skin and subcutaneous tissue disorders) | 1/431 | 7/427
Rash erythematous (Skin and subcutaneous tissue disorders) | 0/431 | 1/427
Rash papular (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Rash pruritic (Skin and subcutaneous tissue disorders) | 1/431 | 0/427
Scar (Skin and subcutaneous tissue disorders) | 0/431 | 1/427
Seborrhoea (Skin and subcutaneous tissue disorders) | 0/431 | 1/427
Skin discolouration (Skin and subcutaneous tissue disorders) | 0/431 | 1/427
Urticaria (Skin and subcutaneous tissue disorders) | 1/431 | 1/427
Myringoplasty (Surgical and medical procedures) | 0/431 | 1/427
Nail operation (Surgical and medical procedures) | 0/431 | 1/427
Tooth extraction (Surgical and medical procedures) | 0/431 | 1/427
Vasectomy (Surgical and medical procedures) | 1/431 | 0/427
Flushing (Vascular disorders) | 0/431 | 1/427
Hot flush (Vascular disorders) | 2/431 | 0/427
Hypertension (Vascular disorders) | 9/431 | 13/427
Systolic hypertension (Vascular disorders) | 1/431 | 0/427
Varicose vein (Vascular disorders) | 0/431 | 1/427

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.